CLINICAL TRIAL: NCT02190266
Title: The Pathogenesis and Genetics of Disseminated or Refractory Coccidioidomycosis
Brief Title: Pathogenesis and Genetics of Disseminated or Refractory Coccidioidomycosis
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140146; 14-I-0146
Record Dates: First submitted 2014-07-12; First posted 2014-07-15 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Coccidioidomycosis
Keywords: Extrapulmonary; Immunodeficiency; Genetics; Infection; Fungal; Natural History
MeSH Terms: conditions — Coccidioidomycosis; Immunologic Deficiency Syndromes; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with confirmed refractory and/or disseminated coccidioidomycosis.

SUMMARY:
Background:

- Coccidioidomycosis is caused by a fungus that grows in the southwest United States and parts of Mexico and South America. This disease is caused by breathing dust containing the fungus. It can lead to serious lung and breathing problems. Rarely, the fungus can infect other body parts. This is called disseminated coccidioidomycosis (DCM). If the fungus stays in the lungs for more than 6 months, it is called refractory coccidioidomycosis (RCM). People with DCM or RCM may have difficulty fighting off infection because of immune system problems. Researchers want to study the immune systems of people with DCM or RCM, to learn more about the disease and the best ways to treat it. They also want to learn more about the types of people that get DCM or RCM and about the fungus that causes it.

Objectives:

- To learn more about DCM and RCM, the fungus that causes these diseases, and the people who get them.

Eligibility:

- People over age 2 with DCM or RCM.

Design:

* Participants will be screened with a review of their medical records.
* At the initial visit, participants will have:
* Medical history and physical exam
* Blood and urine tests. Some blood may be used for genetic testing. The samples will not include participants names. Participants will be notified only if the tests show something urgent about their DCM/RCM. Researchers think this sort of problem will be rare.
* Questionnaire about their DCM/RCM
* Sputum (mucus) collection. They will spit into a cup.
* Participants will have 1 follow-up visit per year. They will have blood tests. They may have other procedures to treat their DCM/RCM.

DETAILED DESCRIPTION:
Coccidioidomycosis (CM) is a fungal disease endemic to the southwestern United States, Northern Mexico, and parts of South America. About 150,000 CM infections are estimated to occur in the United States each year, of which 60% are thought to be asymptomatic. Symptomatic patients typically present with a respiratory syndrome likened to community-acquired pneumonia, while less than 1% of infected individuals are thought to develop refractory disease with or without dissemination. Disseminated infection rarely resolves spontaneously and, although any organ can be affected, tends to involve the skin, lymph nodes, central nervous system and/or the skeletal system. While the risk of disseminated infection is increased in immune suppressed patients, many individuals with no significant prior history have developed debilitating, widespread infection. Causes of refractory and/or disseminated disease in previously healthy individuals have only recently begun to be elucidated, including mutations in the IFNy/IL-12 pathway.

We seek to better characterize the genetic predisposition and treatment of refractory

and/or disseminated coccidioidomycosis. Specifically, we will examine multiple immune factors, characterize the demographics of patients afflicted with this disease, and examine the phylogeny of the infecting organisms. This information will reveal endogenous pathways that might be targets for therapeutic intervention.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for this study, potential participants must meet the following criteria:

1. Age greater than or equal to 2 years old.

   a. Enrollment of pediatric patients who are acutely ill or likely to become acutely ill will be deferred until a time when they are considered medically stable by the PI.
2. Have a positive Coccidioides antigen load or culture proven (a) refractory pulmonary coccidioidomycosis or (b) disseminated coccidioidomycosis.

   1. Refractory pulmonary coccidioidomycosis must have occurred for at least 6 months and includes progressive pulmonary involvement without significant pulmonary cavitation.
   2. Disseminated CM is coccidioidomycosis infection in one or more regions outside of the chest.
3. Agree to undergo genetic testing.
4. Allow their samples to be stored for future research.

EXCLUSION CRITERIA:

1. HIV infection
2. Currently taking more than 20 mg/day of prednisone or undergoing active immunosuppressive therapy in the opinion of the investigator
3. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer s ability to give informed consent.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed refractory and/or disseminated coccidioidomycosis.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-09-02 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Study patients with refractory and/or disseminated coccidioidomycosis in order to identify known and novel immune defects, characterize the demographics of patients afflicted with this disease, follow disease progression in patients, and charact... | Ongoing
  Collecting information on coccidioidomycosis.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Holland, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-I-0146.html